CLINICAL TRIAL: NCT06165172
Title: Early Feasibility Study of the MyoRegulator® for Treatment of ALS
Acronym: ALSEFS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PathMaker Neurosystems Inc. (Industry)
Collaborators: Spaulding Rehabilitation Hospital (Other); Sean M. Healey & AMG Center for ALS (Other); Muscular Dystrophy Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: PMN-004
Record Dates: First submitted 2023-11-28; First posted 2023-12-11 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: amyotrophic lateral sclerosis; neuromodulation; motor neuron hyperexcitability suppression; non-invasive
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Intervention (Experimental): Active treatment with MyoRegulator® device
  Interventions: Device: MyoRegulator®

INTERVENTIONS:
Device: MyoRegulator® — Study participants will receive treatment using the MyoRegulator® device 3 times a week for 2 x 30 minutes per session. The first week of treatment will be followed by a 1-week rest period with no treatments. Treatment sessions will then resume for 4 consecutive weeks, 3 times per week. A follow-up visit will be scheduled 4 weeks after the last treatment session.

SUMMARY:
This is a single-center, single-arm, open-label study aiming to assess the safety and feasibility of the MyoRegulator® device when used to treat individuals with amyotrophic lateral sclerosis (ALS). This study is the first use of the MyoRegulator® device to treat individuals with ALS. The main objective of this study is to confirm that individuals with ALS can tolerate the study treatment regimen without any evidence of serious adverse events related to the use of the device.

The MyoRegulator® device is a non-significant risk (NSR) investigational non-invasive neuromodulation device that uses multi-site direct current (multi-site DCS) stimulation. It has been used in two completed clinical trials evaluating its efficacy to treat post-stroke muscle spasticity and is currently being evaluated in a third trial in this post-stroke population.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS, Lou Gehrig's disease) is a progressive neurodegenerative disease that affects motor neurons in spinal cord and brain. ALS causes motor and cognitive function deficits and eventual death, typically within 2-5 years of diagnosis. There are at least 30,000 ALS patients in the United States and about 5,000 new diagnoses every year according to the Centers for Disease Control (CDC).

Recent research has established important links between ALS and motor neuron hyperexcitability and suggest that motor neuron hyperexcitability is found across different ALS variants.

The multi-site DCS MyoRegulator® treatment is a non-invasive approach to the suppression of motor neuron hyperexcitability based on multi-site direct current stimulation (DCS). Pre-clinical studies show that treatment using multi-site DCS effectively slows disease progression in transgenic mouse models of ALS. This is associated with improved motor function, preservation of motor neurons, and improved animal survival.

This clinical study is a non-significant risk (NSR) investigation using the non-invasive multi-site DCS MyoRegulator® to evaluate the feasibility and safety of treatment with MyoRegulator® in individuals with ALS. The primary endpoint is feasibility and safety. Feasibility will be evaluated by recording and assessing the proportion potential participants who are enrolled from the total number of participants screened for the study, the ease of delivering treatment, the tolerability of study participants to the treatment, and the compliance of study participants with the study schedule and evaluations. Safety will be evaluated by recording the frequency and duration of any adverse events reported by study participants or observed by physical examination during or following treatment and throughout the study duration.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* A clinical diagnosis of ALS as confirmed by medical history
* Willing to forgo botulinum toxin, phenol or alcohol injections, intrathecal baclofen, digitalis, and morphine for the study duration
* Willing to refrain from participation in any other clinical trial for the duration of this study
* Willing to forgo pregnancy for the duration of the study
* Willing and able to give informed consent or have informed consent provided for them by their legal guardian
* Cognitive function sufficient to understand the study and follow instructions (per interview with appropriate clinician)

Exclusion Criteria:

* Study participants who are on permanent assisted ventilation (PAV) defined as >22h of noninvasive or invasive ventilation a day for > 7 consecutive days.
* Implanted intrathecal pump
* Prior botulinum toxin injection(s) within 12 weeks of study enrollment
* Prior phenol or alcohol injections within 6 months of study enrollment
* Presence of potential risk factors for trans-spinal direct current stimulation:
* Damaged skin at the stimulation sites (i.e., skin with ingrown hairs, acne, razor nicks, wounds that have not healed, recent scar tissue, broken skin, etc.)
* Lack of sensory perception at the stimulation sites
* Presence of an electrically, magnetically, or mechanically activated implant (including cardiac pacemaker) or any other electrically sensitive support system with the exception of loop recorders
* Ferrous metal in the path of the current flow (jewelry must be removed during stimulation)
* Past history of epileptic seizures or unexplained spells of loss of consciousness during the previous 36 months
* Any medical condition that would prevent the participant from being able to participate in the clinical outcome measures
* Pregnant females, as determined by a pregnancy test at enrollment (in females of child-bearing potential)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-06-21 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Safety as measured by number of patients with any device-related serious adverse event | Up to 4 weeks following the last treatment
  Safety will be evaluated by recording the frequency, severity, and duration of any adverse events reported by study participants or observed by physical examination during or following treatment and throughout the study duration.
Tolerability as measured by patient's ability to complete the treatments | Up to 4 weeks following the last treatment
  Treatment tolerability will be evaluated by assessing the ease of delivering treatment, the tolerability of study participants to the treatment, and the compliance of study participants with the study schedule and evaluations.

SECONDARY OUTCOMES:
Improvement in Functionality | Up to 4 weeks following the last treatment
  Change in Amyotrophic Lateral Sclerosis Functional Rating Scale - Revised (ALSFRS-R) score following treatment as compared to baseline. The ALSFRS-R measures 12 aspects of physical function, ranging from one's ability to swallow and use utensils to climbing stairs and breathing. Each function is scored from 0 (no ability) to 4 (normal), with a summed total score from 0 (worst) to 48 (best).
Improvement in Activities of Daily Living | Up to 4 weeks following the last treatment
  Change in Rasch Overall ALS Disability Scale (ROADS) score following treatment as compared to baseline.
  The ROADS is a patient-reported outcome measure that assesses overall disability level in people with ALS. The scale contains 28 items, each scored 0 (unable to perform), 1 (can perform but with difficulty), or 2 (normal performance) and a summed total score from 0 (worst) to 56 (best).
Improvement in Quality of Life | Up to 4 weeks following the last treatment
  Change in Amyotrophic Lateral Sclerosis Assessment Questionnaire - 40 (ALSAQ-40) score following treatment as compared to baseline. The ALSAQ-40 consists of 40 questions about how well the patient can perform tasks in 5 areas: physical mobility, activities of daily living and independence, eating and drinking, communication, and emotional reactions. Each task is rated on a five-point scale from 0 = can't do, to 4 = normal ability with a summed total score from 0 (worst) to 40 (best).

CONTACTS AND LOCATIONS:
Overall Officials: J. Leon Morales-Quezada, M.D, Ph.D., Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No